CLINICAL TRIAL: NCT06306157
Title: Low Dose Naltrexone (LDN) Therapy for Complex Regional Pain Syndrome (CRPS): A Feasibility Study
Brief Title: Low Dose Naltrexone Therapy for Complex Regional Pain Syndrome
Acronym: LDN-CRPS
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-0667
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Complex Regional Pain Syndrome; Chronic Pain; Causalgia; Complex Regional Pain Syndrome Type I; Complex Regional Pain Syndrome Type II
Keywords: Chronic pain; Pain management; Drug intervention; CRPS
MeSH Terms: conditions — Complex Regional Pain Syndromes; Chronic Pain; Causalgia; Agnosia | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: This is a feasibility, randomized, placebo-controlled interventional drug study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A quadruple blinded study where the patient, research team, treating clinician, and outcomes assessor are unaware of the randomization results until after study conclusion. The research pharmacy will not be blinded and will be responsible for preparing the medication and securely handing it off to the research assistant according to the pre-approved dispensation plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo sugar capsules (Placebo Comparator): Half of all enrolled patients will be randomized to receive placebo sugar capsules. Neither the patient nor treating physician will be aware of the group in which the patient was randomized into until after study conclusion. All patients will be requested to take the respective daily dose and follow the titration schedule as instructed. All patients enrolled in the study, regardless of their randomization, will have standard of care treatment for CRPS according to their symptoms and the clinical judgment of the treating clinician.
  Interventions: Drug: Placebo sugar capsules
- Low dose naltrexone (Experimental): Half of all enrolled patients will be randomized to receive capsules with the active low dose naltrexone (LDN) ingredient. LDN will be titrated over time to minimize potential side effects, with the initial dose starting at 1.5mg and eventually increasing up to 4.5mg. Neither the patient nor treating physician will be aware of the group in which the patient was randomized into until after study conclusion. All patients will be requested to take the respective daily dose and follow the titration schedule as instructed. All patients enrolled in the study, regardless of their randomization, will have standard of care treatment for CRPS according to their symptoms and the clinical judgment of the treating clinician.
  Interventions: Drug: Low dose naltrexone

INTERVENTIONS:
Drug: Low dose naltrexone — While naltrexone is FDA-approved for treatment of alcohol or opioid addition, this study will be looking at how naltrexone, when dosed very low, may reduce the painful symptoms associated with CRPS. Naltrexone is not FDA-approved for pain management treatment of CRPS at this time, and therefore the study intervention is using the drug in an off-label manner.
  Other Names: LDN
  Arms: Low dose naltrexone
Drug: Placebo sugar capsules — The external appearance of the capsules prepared by the pharmacy will be identical to the LDN capsules. The inactive capsule ingredients will be microcrystalline cellulose (MCC) and Magnesium stearate
  Arms: Placebo sugar capsules

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a rare and often debilitating chronic pain condition whereby individuals may experience extreme sensitivity, discoloration, and swelling of the affected area -- along with numerous other painful symptoms. There are currently a limited number of treatment options available to those suffering with the condition, with various treatments including nerve blocks, neuropathic medications, and desensitization physical therapy modules. There is budding interesting in the role naltrexone, an opiate antagonist, may play in the pain management of CRPS when prescribed in very low doses. This study aims to collect preliminary data on pain scores, symptom severity, and side-effects in patients with Complex Regional Pain Syndrome randomized to receive low dose naltrexone or placebo capsules. Enrollment of 40 patients total will occur over two years from study start to study end. Each patient will be randomized to receive placebo capsules or active low dose naltrexone capsules, with both the patient and treating clinician blind to the randomization. Each patient will be actively enrolled in the study for six months and will take the medication daily at the instructed dose for the respective duration of time. Following the initial visit and study enrollment, the investigators are asking each patient to return for three (3) in-person follow-up office visits. These office visits will occur 1 month after the patient starts the medication, 3 months afterwards, and 6 months afterwards. The final 6-month office visit will mark the conclusion of the patient's active participation in the study.

DETAILED DESCRIPTION:
Naltrexone, an FDA-approved medication since 1984, is classically prescribed in daily doses of at least 50 mg to mediate opiate and alcohol abuse as part of a comprehensive treatment program. By acting as an antagonist in the body, full-strength naltrexone competitively binds to opioid receptors and blocks the effects of opioid-classified drugs, thereby helping to reduce reliance and addiction. In much lower doses (1.5 - 4.5mg per day), naltrexone has been seen to reduce inflammation and nerve pain by instead blocking a different set of receptors involved in cytokine release and uptake. The exact mechanism of naltrexone's ability to decrease inflammation, swelling, and chronic nerve pain is unknown; however further research is being done to discover more. When healthcare providers prescribe naltrexone in these low doses, the medication is referred to as low-dose naltrexone-or LDN.

As of recently, healthcare providers have begun looking at the efficacy of low-dose naltrexone when treating pain caused primarily by the nervous system, referred to as neuropathic pain. Complex Regional Pain Syndrome (CRPS) is a debilitating chronic pain condition caused by dysfunction of or damage to the nervous system. CRPS can be caused by an injury, surgery, or have no obvious cause at all. CRPS typically affects a specific area of the body, such as the hands or feet, and symptoms may include extreme sensitivity, pins-and-needles sensation, color and/or temperature changes, swelling, and stinging. One treatment route commonly prescribed for CRPS is an anti-neuropathic medication regime of Gabapentin or Pregabalin-medications prescribed to specifically ease nerve-related pain. Targeted nerve blocks and epidural injections are other common treatments physiatrists and pain providers will perform for CRPS patients, often in conjunction with medication and physical therapy for a comprehensive pain management plan. However, for those who cannot take anti-neuropathic medications and are hesitant to pursue more invasive routes like nerve blocks or spinal cord stimulations, there is a lack of available treatment options which makes pain management uncertain and inconsistent. In an effort to diversify available treatments, there is a budding interest in the role that low-dose naltrexone may play in reducing chronic pain associated with CRPS.

There is currently only one other low-dose naltrexone study being conducted with Complex Regional Pain Syndrome patients as the primary study population. Dr. Sean Mackey is leading this study through the Stanford Division of Pain Medicine, and the study is still in the process of enrolling eligible patients. Published case studies demonstrate the promising nature of the drug in a multi-modal treatment course and suggest that more extensive research on the effectiveness of low-dose naltrexone would be beneficial. When physicians wish to incorporate LDN into the treatment course for a CRPS patient, they have additional barriers to cross because naltrexone is FDA-approved only for alcohol and opioid-use disorders. The lack of FDA-approval for naltrexone in CRPS treatment creates limited accessibility to the drug, the need for compounding pharmacy involvement, and a lack of education surrounding low-dose naltrexone in the CRPS and chronic pain community. Conducting controlled clinical trials and thereby learning more about the efficacy of low-dose naltrexone and possible side effects or adverse reactions would help establish LDN as another treatment possibility for frustrated patients dealing with this chronic pain syndrome.

Our feasibility study has two purposes: to evaluate the potential of LDN as CRPS pain management, and to evaluate whether such a long-term interventional drug study can be conducted at the Hospital for Special Surgery (HSS). Not only will the investigators be collecting pain scores over time to better understand whether LDN may help improve pain and symptom severity, but the investigators will also be collecting information regarding how many patients enroll, how many patients remain enrolled during the duration of the study, why patients may un-enroll, and how compliant patients are with taking the daily study medication. This study will be requesting that each enrolled patient take a medication every day for 6 months, consistently attend office visits when requested, and take record of how often they miss a dose. To date and to our knowledge, no similar study requiring such extensive participation and long-term medication consumption has been conducted at HSS-whether in the main hospital or through an outpatient clinic. In order to expand on the knowledge base HSS has developed regarding its chronic pain patient population, long-term research utilizing placebo and study medication is essential. Prior to conducting larger-scale interventional drug studies, it is imperative that the workflow is streamlined and established protocols are in place. Aside from looking into the LDN-CRPS relationship, the main purpose of this feasibility study is to develop an infrastructure to demonstrate that interventional drug studies of this magnitude are possible at HSS, establish novel protocols and standard operating procedures, and gauge the receptiveness of chronic pain patients to studies of this kind at HSS.

Over the course of two years, a total of 40 patients recently diagnosed with CRPS at the 75th St HSS outpatient location will be enrolled and randomized to receive either capsules with the active low-dose naltrexone medication, or placebo capsules which do not contain any active ingredient. The study medication will be supplied to study patients in addition to any standard CRPS therapies, including physical therapy, medication management, and interventional therapies. Enrolled patients will take the medication every day for a total of 6 months and will attend standard of care office visits after 1 month, after 3 months, and after 6 months. Before each visit, patients will be asked to record their daily average pain for one week leading up to the visit. In between office visits, a study team member will be calling the patients to record medication consumption compliance, pain scores, questionnaire responses, adverse reactions, and any side effects. Questionnaires will include PROMIS-10, S-LANSS, and an NRS screening. A study team member will also be calling patients as a reminder to record in their 7-day pain diary when necessary. A major component of the study protocol is the titration schedule-a schedule that defines how the drug dosage will increase over time-which Dr. Semih Gungor, the principal physician investigator, has already established at his clinic. While it is subject to change depending on the patient's CRPS symptom progression and medication-related side effects, the titration schedule built into the study protocol will be starting at 1.5mg during the 1st month, increasing to 3mg the 2nd month, and finally up to 4.5mg the 3rd month and beyond. The purpose of this titration schedule is to limit the side effects a patient may feel when starting on naltrexone and to gradually introduce them to the drug to facilitate a long-term treatment.

Through the enrollment of study patients and successful dispensation of daily medication over a 6-month time period, our study aims to collect preliminary data on pain scores, symptom severity, and side-effects in patients randomized to LDN vs. placebo, as well as determine the feasibility of conducting a long-term interventional drug study-with the goal of expanding future research opportunities at HSS and supplementing treatment courses for those struggling with this often debilitating chronic pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years old
* Meeting CRPS diagnostic criteria using the Budapest Clinical Diagnostic Criteria
* CRPS patients with severe pain (NRS>3) that affects their daily life.
* CRPS patients with pain and other symptoms for more than 3 months.

Exclusion Criteria:

* Patients with suspected disc herniation, spinal stenosis, myelopathy, and suspected radiculopathy in detailed examinations and examinations (MRI, CT).
* Systemic or local infection
* Malignancy
* Current or planned pregnancy within the study period.
* Uncontrolled medical and psychiatric condition
* Patients with known liver issues, including but not limited to end-stage liver disease, severe cirrhosis or an acute hepatic state.
* Patients who are currently using opioid drugs
* Patients who are currently using alcohol or considering using alcohol during the study period.
* Allergy to naltrexone or naloxone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of study patients enrolled | Within 2 years of study start
  Enrollment of 40 patients within two years is the target (i.e. enrollment of 1-2 patients a month). If 1-2 patients a month is not being met within first 6 months, an invitation to other chronic pain co-investigators with high volume CRPS will be considered. Because this is a feasibility study, determining whether 40 patients can be enrolled with the current inclusion and exclusion criteria within a specified time frame is an essential step in ensuring such a long-term outpatient study can be conducted.
Number of study patients randomized | At initial time of enrollment
  Measured as completed or not. Quadruple blinded randomization of each study patient to one of the two treatment arms after enrollment and before medication dispensation will be deemed successful. Because this is a feasibility study, determining whether 40 patients can be blindly randomized to a group according to the protocol is an essential step in ensuring such a long-term drug study can be conducted.
Number of study patients who received the study medication | At initial time of enrollment and at 3 months.
  Dispensation of medication to all enrolled study patients at point of enrollment and at 3 months will be considered successful. If deemed necessary, dispensation can occur at time points other than the two previously defined and will still be considered successful if patient receives medication on time. Because this is a feasibility study implementing a long-term interventional drug treatment, it is essential that the investigators are measuring whether medication dispensation is occurring on time and according to the protocol.

SECONDARY OUTCOMES:
Incidence of side effects/adverse events | 1, 3, and 6 months
  Side effects or adverse events, including sleep disturbances, mild headaches, mild agitation, and nausea. Study patients are encouraged to contact the study team outside of study visits to report side effects/adverse events as they arise throughout course of the study, but the outcome is formally assessed at the below time points.
Average NRS pain | Baseline, 1, 3, and 6 months.
  Pain measured using numerical rating scale (NRS) from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable. NRS at baseline will be self-reported average at time of visit; NRS at 1, 3, and 6 months will be 7-day average leading up to those timepoints, collected via a patient diary.
CRPS symptom severity | Baseline, 1, 3, and 6 months.
  CRPS symptom severity score (CSS) based on the Budapest Criteria which measures the severity of CRPS over time on a scale from 0-16 via the presence or absence of 8 specific symptoms and 8 specific signs. CSS will be measured at the respective in-person office visit.
PROMIS-10 score | Baseline, 1, 3, and 6 months
  The PROMIS-10 (Patient-Reported Outcomes Measurement Information System) score has two components, a physical score and a mental score, and is captured via a self-administered questionnaire with the purpose of assessing the patient's health-related quality of life. PROMIS-10 assessments are scored using T-score metrics and are calculated based on patient responses to the 10-item questionnaire. For the physical PROMIS-10 score, the lowest possible is 16.2 and the highest possible is 67.7. For the mental score, the lowest is 21.2 and the highest is 67.6. The higher a patient scores in each category, the greater their respective health is. A physical and mental T-score above 58 and 56, respectively, is rated "Excellent", whereas a physical and mental T-score below 35 and 29 is rated "Poor".
S-LANSS score | Baseline, 1, 3, and 6 months
  S-LANSS (Self-Administered Leeds Assessment of Neuropathic Symptoms and Signs) score which aims to characterize the extent to which pain is neuropathic in origin on a scale from 0-24. The score is captured via a 7-item self-administered questionnaire.
Blinding assessment | 1, 3, and 6 months
  Patients are asked which treatment they think they received. The correctness of their guesses is then measured using the bang-blinding index to see if patients were able to accurately guess which treatment they received. It is measured on a scale of -1 to 1. Scores closer to 0 indicate better blinding, or patients not being able to guess their treatment.

OTHER OUTCOMES:
Enrollment rate | At study completion (approximately 2 years after study initiation)
  Monitored over the course of the study and measured by number of eligible patients who enroll/total number of eligible patients.
Study medication compliance | 1, 3, and 6 months
  Patient-reported and patient-prompted qualitative measure of the extent to which a patient complied with the study medication regimen, including taking the daily medication at the appropriate dose. Recorded at office visits and via daily patient diary. At the below time points, medication compliance during the previous time period is being recorded. (i.e During the 3-month office visit, the patient will be asked "Have you missed taking your daily medication on any day since the 1-month visit").
Reasons for study medication non-compliance | 1, 3, and 6 months
  Reasons for missing a dose, including side effect(s), forgetting, unsuccessful medication dispensation, or being away from medication (i.e. vacation). Recorded at office visits and via patient diary. At the below time points, reasons for medication non-compliance during the previous time period is being recorded. (i.e During the 3-month office visit if the patient reports missing the medication at least once, they will be asked for the corresponding reason).
Drop-out rate | 1, 3, and 6 months
  Whether a patient prematurely withdrew due to any reason from the study before reaching the final 6-month office visit, measured as "Yes, patient dropped out of the study," or "No, patient did not drop out". The investigators will consider the study as having a low-drop rate at its conclusion if 80% of patients are retained through the 6-month follow-up. If the patient contacts the study team to drop out in between the time points listed below, the data will be recorded on the form corresponding to the next office visit. (i.e. if the patient contacts the study team on day 70 and requests to drop out, the team will record the subsequent information in the 3-month office visit form, recording the exact day the patient dropped out. Otherwise, the data will be collected at the time points listed below).
Reasons for drop-out | 1, 3, and 6 months
  Reasons for a patient dropping out of the study early, including whether it was a self-withdrawal or study team-withdrawal. Reasons include compliance issue, undesirable side effect, lost to follow up, medication dispensation logistic issue, or major contraindication to the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Gungor, M.D., Principal Investigator — Hospital for Special Surgery, New York; Alexandra Sideris, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: For researchers who provide a methodologically sound proposal and analyses to achieve aims in the approved proposal. Proposals should be directed to siderisa@hss.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Toljan K, Vrooman B. Low-Dose Naltrexone (LDN)-Review of Therapeutic Utilization. Med Sci (Basel). 2018 Sep 21;6(4):82. doi: 10.3390/medsci6040082. PMID 30248938
- [Background] Chopra P, Cooper MS. Treatment of Complex Regional Pain Syndrome (CRPS) using low dose naltrexone (LDN). J Neuroimmune Pharmacol. 2013 Jun;8(3):470-6. doi: 10.1007/s11481-013-9451-y. Epub 2013 Apr 2. PMID 23546884